CLINICAL TRIAL: NCT01407016
Title: A Phase 1, Open Study To Assess The Safety, Tolerability And Pharmacokinetics Of Metronidazole Following Single And Multiple Intravenous Infusion In Healthy Japanese Adult Subjects
Brief Title: A Study To Assess The Safety, Tolerability And Pharmacokinetics Of Metronidazole Injection In Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6831006
Record Dates: First submitted 2011-07-20; First posted 2011-08-01 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Infection
Keywords: metronidazole infusion
MeSH Terms: conditions — Infections

ARMS (1):
- 1.0 (Experimental)
  Interventions: Drug: metronidazole IV 500 mg

INTERVENTIONS:
Drug: metronidazole IV 500 mg — On Day 1, subjects will receive a single dose of 500 mg metronidazole by intravenous infusion over 20 minutes. On Day 3 to Day 7, subjects will receive multiple doses of 500 mg metronidazole by intravenous infusion over 20 minutes 4 times a day (every 6 hours) for 5 days.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of metronidazole following single and multiple intravenous infusion in healthy Japanese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and/or female subjects.

Exclusion Criteria:

* Subject with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Subject with history of regular alcohol consumption exceeding 7 drink/week for females or 14 drinks/week for males [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months of screening.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma metronidazole pharmacokinetic parameters for single dose:Cmax | Day 1 to Day 3
Plasma metronidazole pharmacokinetic parameters for single dose:AUClast | Day 1 to Day 3
Plasma metronidazole pharmacokinetic parameters for single dose:AUC0-6 | Day 1 to Day 3
Plasma metronidazole pharmacokinetic parameters for single dose:Tmax | Day 1 to Day 3
Plasma metronidazole pharmacokinetic parameters for multiple dose:Ctrough | prior to Day 3 and Day 6-8 morning dose and 6 hours post morning dose on Day 8
Plasma metronidazole pharmacokinetic parameters for multiple dose:Cmax | Day 8 to Day 9
Plasma metronidazole pharmacokinetic parameters for multiple dose:AUC0-6 | Day 8 to Day 9
Plasma metronidazole pharmacokinetic parameters for multiple dose:Tmax | Day 8 to Day 9
Plasma metronidazole pharmacokinetic parameters for multiple dose:CL | Day 8 to Day 9

SECONDARY OUTCOMES:
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for single dose: Cmax | Day 1 to Day 3
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for single dose: AUClast | Day 1 to Day 3
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for single dose: AUC0-6 | Day 1 to Day 3
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for single dose: Tmax | Day 1 to Day 3
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for multiple dose: Ctrough | prior to Day 3 and Day 6-8 morning dose and 6 hours post morning dose on Day 8
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for multiple dose: Cmax | Day 8 to Day 9
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for multiple dose: AUC0-6 | Day 8 to Day 9
Plasma 1-(2-hydroxyethyl)-2-hydroxymethyl-5-nitroimidazole pharmacokinetic parameters for multiple dose: Tmax | Day 8 to Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6831006&StudyName=A%20Study%20To%20Assess%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20Metronidazole%20Injection%20In%20Healthy%20Japanese%20Subjects